CLINICAL TRIAL: NCT03865277
Title: Individualized Radiation Dose Prescription in HNSCC Based on F-MISO-PET Hypoxia-Imaging: Multi-center, Randomized Phase-II-trial
Brief Title: Individualized Radiation Dose Prescription in HNSCC Based on F-MISO-PET Hypoxia-Imaging
Acronym: INDIRA-MISO
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Mechthild Krause, Director of the Department of Radiotherapy and Radiation Oncology, Technische Universität Dresden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STR-INDIRA-MISO-2014
Record Dates: First submitted 2019-02-26; First posted 2019-03-06 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Head and neck cancer; radiochemotherapy; HPV
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- standard radiochemotherapy, hypoxic (Other): HPV (-), hypoxic in 18F-MISO PET after 2 weeks of radiochemotherapy, randomized to standard radiation dose, 70 Gy standard radiochemotherapy
  Interventions: Radiation: standard radiochemotherapy
- dose-escalated radiochemotherapy, hypoxic (Experimental): HPV (-), hypoxic in 18F-MISO PET after 2 weeks of radiochemotherapy, randomized to escalated radiation dose, 77 Gy radiochemotherapy
  Interventions: Radiation: dose-escalated radiochemotherapy
- escalated radiochemoth., carbon boost, hypoxic (Experimental): HPV (-), hypoxic in 18F-MISO PET after 2 weeks of radiochemotherapy, non-randomised arm (only possible in the trial center Heidelberg), 77 Gy radiochemotherapy (boost with carbon)
  Interventions: Radiation: dose-escalated radiochemotherapy with carbon ion boost
- standard radiochemotherapy, oxic (Other): HPV (-), oxic in 18F-MISO PET after 2 weeks of radiochemotherapy, 70 Gy standard radiochemotherapy
  Interventions: Radiation: standard radiochemotherapy
- standard radiochemotherapy (70 Gy) (Other): HPV (+), HPV positive patients will get the same imaging and clinical examinations as HPV negative patients. This measure is necessary to further elucidate the prognostic role of hypoxia and HPV status and their correlation, the information will be important for consecutive clinical trials. 70 Gy standard radiochemotherapy.
  Interventions: Radiation: standard radiochemotherapy

INTERVENTIONS:
Radiation: dose-escalated radiochemotherapy — Patients will receive simultaneous radiochemotherapy, however the simultaneous chemotherapy is standard and not part of the evaluation in this trial. Present standard chemotherapy is cisplatinum 40 mg/m²/week (chemotherapy over the whole course of radiotherapy).
  Radiotherapy is applied to doses of 54 Gy(RBE)/ 1.8 Gy(RBE) per fraction to the adjuvant region, 70 Gy(RBE)/ 2 Gy(RBE) per fraction to the tumor and involved lymphonodes and, if "hypoxic" and randomized to the intervention arm, 77 Gy(RBE)/ 2.2 Gy(RBE) per fraction to the primary tumor and lymphonode metastases > 2 cm.
  Radiotherapy is always applied with 5 fractions per week.
  Arms: dose-escalated radiochemotherapy, hypoxic
Radiation: dose-escalated radiochemotherapy with carbon ion boost — Patients will receive simultaneous radiochemotherapy, however the simultaneous chemotherapy is standard and not part of the evaluation in this trial.
  Radiotherapy is applied to doses of 54 Gy(RBE)/ 1.8 Gy(RBE) per fraction to the adjuvant region, 70 Gy(RBE)/ 2 Gy(RBE) per fraction to the tumor and involved lymphonodes and, if "hypoxic" and treated in the study site Heidelberg, 77 Gy(RBE)/ 2.2 Gy(RBE) per fraction to the primary tumor and lymphonode metastases > 2 cm using a carbon ion boost.
  Radiotherapy is always applied with 5 fractions per week.
  Arms: escalated radiochemoth., carbon boost, hypoxic
Radiation: standard radiochemotherapy — Patients will receive simultaneous radiochemotherapy, however the simultaneous chemotherapy is standard and not part of the evaluation in this trial. Present standard chemotherapy is cisplatinum 40 mg/m²/week (chemotherapy over the whole course of radiotherapy).
  Radiotherapy is applied to doses of 54 Gy(RBE)/ 1.8 Gy(RBE) per fraction to the adjuvant region and 70 Gy(RBE)/ 2 Gy(RBE) per fraction to the tumor and involved lymphonodes.
  Radiotherapy is always applied with 5 fractions per week.
  Arms: standard radiochemotherapy (70 Gy); standard radiochemotherapy, hypoxic; standard radiochemotherapy, oxic

SUMMARY:
The trial evaluates the value of radiation dose escalation based on Hypoxia detection by 18F_misonidazole Positron Emission Tomography (18F-MISO-PET) for primary radiochemotherapy of head and neck squamous cell carcinoma. Patients negative for human papillomavirus (HPV) and with hypoxic tumours after 2 weeks of radiochemotherapy are randomized to completion of standard radiochemotherapy or radiochemotherapy with escalated radiation dose. An additional interventional arm includes a carbon ion boost. HPV positive tumours can be included in a control arm. Primary endpoint is local tumour control 2 years after radiochemotherapy.

DETAILED DESCRIPTION:
Previous preclinical data and a prospective validated patient cohort have shown that patients with head and neck squamous cell carcinoma, whose tumours are hypoxic after 2 weeks of primary radiochmeotherapy, have a significantly lower chance of locoregional tumour control. The multi-center trial evaluates the value of radiation dose escalation based on hypoxia detection by 18F_misonidazole Positron Emission Tomography (18F-MISO-PET) for primary radiochemotherapy of head and neck squamous cell carcinoma. Patients negative for human papillomavirus (HPV) and with hypoxic tumours after 2 weeks of radiochemotherapy are randomized to completion of standard radiochemotherapy (70 Gy) or radiochemotherapy with escalated radiation dose (77 Gy). An additional interventional arm includes a carbon ion boost to 77 Gy. HPV positive tumours can be included in a control arm. Primary endpoint is local tumour control 2 years after radiochemotherapy. Secondary endpoints include acute and late toxicity (CTCAE 5.0), regional tumor control, overall survival, disease free survival, distant metastases, kinetics analysis of dynamic FMISO-PET scans, Quality of life (QoL). The hypothesis is that local tumour control 2 years after radiochemotherapy is higher in the dose escalated compared to the control arm.

ELIGIBILITY:
Inclusion Criteria:

* Age: older than 18 years
* WHO (ECOG) performance status 0-2
* Histological proven HNSCC
* HPV negative tumors or HPV positive tumors
* Stage III, IVA or IVB HNSCC according to UICC and AJCC guidelines
* Tumor classified as irresectable or patient inoperable or patient refused surgery
* Tumor extension and localization suitable for radiochemotherapy with curative intent
* Simultaneous standard chemotherapy with cisplatin applicable (no contra-indications)
* Dental examination and -treatment before start of therapy
* For women with childbearing potential and men in reproductive ages adequate contraception.
* Ability of subject to understand character and individual consequences of the clinical trial
* Written informed consent (must be available before enrolment in the trial)

Exclusion Criteria:

* Refusal of the patients to take part in the trial
* Presence of distant metastases (UICC stage IVC)
* Previous radiotherapy in the head and neck region
* Second malignancy that is likely to require treatment during the trial intervention or follow-up period or that, in the opinion of the physician, has a considerable risk of recurrence or metastases within the follow-up period
* Serious disease or medical condition with life expectancy of less than one year
* Participation in competing interventional trial on cancer treatment
* Patients who are not suitable for radiochemotherapy
* Pregnant or lactating women
* Patients not able to understand the character and individual consequences of the trial
* Nasopharyngeal Carcinomas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
local tumour control | Local tumor control 2 years after end of treatment
  Local tumour control (MRI, CT, PET or clinical evaluation) in the randomized dose-escalated arm compared to the randomized non dose escalated arm (arms 1 and 2).

SECONDARY OUTCOMES:
late toxicity | 30 days to 2 years after radiochemotherapy
  late toxicity based on CTCAE 5.0
survival | 2 years after radiochemotherapy
  Overall survival
quality of life EORTC QLQ-C30/HN-35 | regularly up to 2 years after radiochemotherapy
  EORTC-QLQ (C30 and HN-35) Sheets (General for tumour diseases and specific for head and neck cancer)
acute toxicity | during treatment and up to 30 days after radiochemotherapy
  acute toxicity based on CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Mechthild Krause, Prof., Study Chair — University of Technology, University Hospital Carl Gustav Carus, Department of Radiation Therapy and Radiation Oncology, German Consortium for Translational Cancer Research (DKTK)
Locations (8):
- Germany (8):
  - Medical Faculty, Albert-Ludwigs-Universität Freiburg, Department of Radiation Oncology, Freiburg im Breisgau, Baden-Wurttemberg
  - Department of Radiation Oncology Heidelberg University Medical School, Heidelberg, Baden-Wurttemberg
  - Universitätsmedizin Mannheim, Klinik für Strahlentherapie und Radioonkologie, Mannheim, Baden-Wurttemberg
  - Uniklinikum Wuerzburg, Würzburg, Bavaria
  - Mechthild Krause, Dresden, Saxony
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Charité University Hospital, Berlin
  - Ludwig-Maximilian-Universität, Klinikum Großhadern, München

IPD SHARING:
Plan to Share IPD: Undecided